CLINICAL TRIAL: NCT03540004
Title: A Prospective, Single-blind, Multi-center Clinical Study Evaluating the Use of MolecuLight i:X as an Adjunctive Fluorescence Imaging Tool to Clinical Signs and Symptoms for the Identification of Bacteria-containing Wounds.
Brief Title: Evaluation of MolecuLight i:X as an Adjunctive Fluorescence Imaging Tool to Clinical Signs and Symptoms for the Identification of Bacteria-containing Wounds
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MolecuLight Inc. (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Other Study IDs: 18-001
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Soft tissue core biopsies will be obtained from patients with wounds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: MolecuLight i:X Imaging Device — The i:X Imaging Device uses built-in light-emitting diodes (LEDs) emitting 405 nm violet excitation light to illuminate the wound during fluorescence imaging in (FL-Mode). The light excites biological components of the wound and surrounding tissues. Non-biological components may also fluoresce although their presence in wounds is less common, provided the wound has been cleaned following standard care protocols. The resulting wound fluorescence wavelengths emitted are typically between 420 - 700 nm in the visible wavelength spectrum. In FL-mode, a customized fluorescence emission filter, which is mechanically placed in front of the built in imaging sensor and allows real-time capture of wound, limits the visualization of fluorescence to wavelengths between 500-545 nm, which typically appears green in color, and 600-665 nm, which typically appears red in color.

SUMMARY:
This is a non-randomized evaluation for which 160 adult patients will be imaged at outpatient wound care clinics who present with a wound of unknown infection diagnostic status and are receiving standard treatment. The MolecuLight i:X Imaging Device will be used as an adjunctive tool in the assessment of the wound and may be used to guide the targeted sampling of a wound (using a conventional punch biopsy method).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects presenting at an advanced outpatient wound care clinic with wound(s) (e.g. DFU, VLU, PU, SSI)
* 18 years or older

Exclusion Criteria:

* Treatment with an investigational drug within 1 month before study enrolment
* Subjects with recent (<30 days) biopsy of target wound
* Subjects with wounds that cannot be completely imaged by study device due to anatomic location
* Inability to consent
* Any contra-indication to routine wound care and/or monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects presenting at an advanced outpatient wound care clinic with wound(s) (e.g. DFU, VLU, PU, SSI)
Sampling Method: Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of identifying wounds with moderate/heavy bacterial load as measured by sensitivity and specificity. | 1 year
  Superiority in sensitivity of clinical signs and symptoms (CSS) and fluorescence imaging using MolecuLight i:X (CSS + i:X) vs. CSS alone to identify wounds with moderate/heavy bacterial load
  Non-Inferiority of specificity of CSS and fluorescence imaging using MolecuLight i:X (CSS + i:X) vs. CSS alone with region of indifference of 10% to identify wounds with moderate/heavy bacterial load

SECONDARY OUTCOMES:
Estimation of sensitivity and specificity of MolecuLight i:X alone | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tomas E Serena, MD, Principal Investigator — Serena Group Research Institute
Locations (14):
- United States (14):
  - New Hope Podiatry Group, Los Angeles, California
  - Royal Research Group, Pembroke Pines, Florida
  - Saint Mary's Center for Wound Healing, Athens, Georgia
  - The Wound Treatment Center at Opelousas General Health System, Opelousas, Louisiana
  - Cleveland Foot and Ankle Clinic, Cleveland, Ohio
  - The Heal Clinic, Tulsa, Oklahoma
  - Foot and Ankle Center, Bryn Mawr, Pennsylvania
  - Saint Vincent Health Center, Erie, Pennsylvania
  - The Foot and Ankle Wellness Center of Western Pennsylvania, Ford City, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - Serena Group Research Institute, Pittsburgh, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania
  - El Campo Memorial Hospital, El Campo, Texas
  - Texas Gulf Coast Medical Group, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson J, Johnson AR Jr, Andersen CA, Kelso MR, Oropallo AR, Serena TE. Skin Pigmentation Impacts the Clinical Diagnosis of Wound Infection: Imaging of Bacterial Burden to Overcome Diagnostic Limitations. J Racial Ethn Health Disparities. 2024 Apr;11(2):1045-1055. doi: 10.1007/s40615-023-01584-8. Epub 2023 Apr 11. PMID 37039975
- [Derived] Serena TE, Gould L, Ousey K, Kirsner RS. Reliance on Clinical Signs and Symptoms Assessment Leads to Misuse of Antimicrobials: Post hoc Analysis of 350 Chronic Wounds. Adv Wound Care (New Rochelle). 2022 Dec;11(12):639-649. doi: 10.1089/wound.2021.0146. Epub 2021 Dec 3. PMID 34714159